CLINICAL TRIAL: NCT02641405
Title: Efficacy of Proprioceptive Focal Stimulation (EQUISTASI) on Gait Parameters in Parkinson. Italian Multicentric Study
Acronym: PAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Collaborators: Istituto Auxologico Italiano (Other); IRCCS National Neurological Institute "C. Mondino" Foundation (Other); Ospedale S. Raffaele Arcangelo, Fatebenefratelli (Other); University of Genova (Other); IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Antonella Peppe, MD, PhD, I.R.C.C.S. Fondazione Santa Lucia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CE/PROG.478
Record Dates: First submitted 2015-12-03; First posted 2015-12-29 (Estimated); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Parkinson Disease; Gait, Shuffling; Effects of Vibration
Keywords: Gait analysis; Proprioceptive focal stimulation; Parkinson
MeSH Terms: conditions — Parkinson Disease; Gait Disorders, Neurologic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Equistasi (Experimental): Equistasi is a nanotechnology for proprioceptive focal stimulation. Every patient will receive three patches to be placed at C7 and at the gastrocnemial junction of both legs.
  Interventions: Device: Equistasi
- Placebo (Placebo Comparator): Inactive Equistasi will be given to every patient in the form of three patches to be placed at C7 and at the gastrocnemial junction of both legs.
  Interventions: Device: Inactive Equistasi

INTERVENTIONS:
Device: Equistasi — Equistasi is a nanotechnology for proprioceptive focal stimulation. Every patient will receive three patches to be placed at C7 and at the gastrocnemial junction of both legs.
  Arms: Equistasi
Device: Inactive Equistasi — Inactive Equistasi will be given to every patient in the form of three patches to be placed at C7 and at the gastrocnemial junction of both legs.
  Arms: Placebo

SUMMARY:
It's already known the efficacy of Gait Analysis (GA) on evaluating gait modification on Parkinson's Disease (PD) Patients (1). On the other hand Proprioceptive Focal Stimulation seems be useful in symptoms amelioration in several neurological disease. Few studies have been performed in Parkinson's disease. A total of 126 patients suffering from PD will be recruited in 6 italian neurological centers. The study will be a cross-over multicenter study with the randomization of the sequence. The patients will be randomly assigned to 2 groups receiving for 8 weeks either the Equistasi medical device, or an equivalent placebo. Gait analysis will be recorded in each patient at the beginning and at the end of the treatment assigned. After 4 weeks of wash-out, the treatment will be crossed and a new gait analysis recording will be performed. Finally a last recording will be taken at the end of the last 8 weeks. Secondary outcome will be the MDS-UPDRS (Movement Disorder Society - Unified Parkinson Disease Rating Scale), PDQ-39 (Parkinson Disease 39 Questionnaire ), ABC (Activity Specific Balance Confidence Scale).

ELIGIBILITY:
Inclusion Criteria:

* Patient with rigid-acinetic bilateral PD form
* At least 4 years of disease history
* H&Y between 2-3
* Stable drug therapy response without any change performed in the 3 months before the study.
* Presence of freezing (FOG) and of postural instability not responding to parkinsonian therapy.
* MMSE>24/30 (Mini-Mental State Examination)

Exclusion Criteria:

* Systemic illness
* Presence of cardiac pacemaker
* Presence of deep brain stimulation
* Presence of severe dysautonomia with marked hypotension
* Obsessive-Compulsive disorder (OCD)
* Major depression
* Dementia
* History or active neoplasia
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Changes in Spatio-Temporal gait variables at 20 weeks | 20 weeks

SECONDARY OUTCOMES:
Changes in the Movement Disorder Society - Unified Parkinson Disease Rating Scale (MDS-UPDRS) - at 20 weeks | 20 weeks
Changes in the Parkinson Disease 39 Questionnaire (PDQ-39) at 20 weeks | 20 weeks
Changes in the Activity Specific Balance Confidence Scale (ABC scale) at 20 weeks | 20 weeks

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - IRCCS Santa Lucia, Rome, Lazio
  - IRCCS National Neurological Institute "C. Mondino" Foundation, Pavia, PV
  - Istituto Auxologico Italiano, Oggebbio, Verbano-Cusio-Ossola
  - IRCCS San Raffaele, Cassino
  - University of Genova, Genova
  - Ospedale S. Raffaele Arcangelo, Fatebenefratelli, Venezia